CLINICAL TRIAL: NCT06012032
Title: Application in Rehabilitation of BHOHB SPINAL-METER and CervicalMeter for the Assessment of Posture in Patients With Dysmorphisms and Paramorphisms of the Spine
Brief Title: Application of BHOHB SPINAL-METER and CervicalMeter for Posture Assessment
Acronym: BHOHB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 4381
Record Dates: First submitted 2023-03-10; First posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Parkinson Disease; Osteoporosis; Scoliosis; Postural; Defect
MeSH Terms: conditions — Parkinson Disease; Osteoporosis; Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The postural observation of the patient has an important role for the evaluation and monitoring of orthopedic and neurological degenerative pathologies. The study of the effects of rehabilitation in the treatment of postural alterations depends on the validity, sensitivity and specificity of the tool used.

The radiographic evaluation of the spine in the standard anteroposterior and lateral projections is the gold standard and provides a standardized and objective measure of the dysmorphisms and paramorphisms of the spine, although it requires exposure to X-rays and with costs of the method especially in the need to repeat the radiological examination in time.

Non-radiological tools for postural assessment have been proposed in the literature, with uncertain judgments by the various authors regarding their validity and reliability, due to the heterogeneity and poor quality of the studies in this regard.

The aim of this study is to evaluate the effectiveness of a new posture analysis methodology (BHOHB SPINAL-METER ® and CervicalMeter®) in measuring spine dysmorphisms and paramorphisms in adult patients affected by orthopedic and neurological degenerative pathologies, who carry out rehabilitation at the Policlinico Gemelli Foundation (FPG) Hospitalization and Rehabilitation Services clinic. In particular, the correspondence of radiological and clinical data with the reports obtained from the "BHOHB SPINAL-METER ® and CervicalMeter®" will be considered and the relationship between the data obtained with the two methods and the characteristics of pain, disability, balance and quality of life will be observed of patients suffering from orthopedic and neurological disease with dysmorphisms and paramorphisms of the spine, belonging to the rehabilitation clinic who agree to participate in the study.

DETAILED DESCRIPTION:
Setting: outpatients ward, UOSA( "Unità operativa semplice ambulatoriale" simple outpatient operating unit) Rehabilitation Service Hospitalization and FPG Rehabilitation Services.

Duration of the study: 1 year

Goals:

Primary endpoint: evaluation of the correlation of radiological and clinical reports with those obtained from the device under study; in particular, the measurement of the radiological Cobb angle (from standard X-ray in orthostatism, on a single plate in the anteroposterior projection) of the patient will be correlated with that evaluated with the BHOHB SPINAL-METER® and CervicalMeter® Secondary end point: evaluation of the effects of postural alteration measured radiologically and with the "BHOHB SPINAL-METER ® and CervicalMeter®" on static and dynamic balance, on spine pain and on the quality of life of patients, evaluated respectively with the measures Berg Balance scale, Tinetti Gait Evaluation, NRS (Numeric rating Scale) and with stabilometric examination, which are performed routinely in outpatient visits.

Calculation of the sample size: Based on the current literature on the results obtained via RX and on the data of the new instrument held by the investigators, in order to estimate a Pearson correlation coefficient equal to 0.90, with a width of the interval of 0.10 and a bilateral confidence interval of 95%, it is considered necessary to enroll a minimum number of patients equal to 62.

Statistical analysis: Qualitative variables will be described through absolute frequencies and percentages, while quantitative variables as mean and standard deviation or median and interquartile range according to their distribution, which will be tested through the Shapiro-Wilk test.

The evaluation of the degree of correlation between the measurement of the radiological Cobb angle of the patient with that evaluated with the BHOHB SPINAL-METER ® and CervicalMeter® will be performed by calculating the Pearson correlation coefficient, and further exemplified by suitable scatter plots.

The effects of postural alteration measured radiologically and with the BHOHB SPINAL-METER ® and CervicalMeter®, on static and dynamic balance, spine pain and patients' quality of life will be analyzed through univariate and multivariate linear regression models.

A p-value <0.05 will be considered statistically significant. The statistical analyzes will be performed using the STATA 16 software.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged > 18 years
* MMSE >23
* Subjects affected by orthopedic and neurological degenerative pathologies and with dysmorphisms or paramorphisms of the spine, capable of maintaining an upright position and ambulating without aids.
* Signature of the informed consent

Exclusion Criteria:

* Psychiatric pathologies,
* Cognitive impairment (MMSE<23),
* Inability to stand and walk.
* Failure to sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients affected by dysmorphisms and paramorphisms of the spine due to degenerative orthopedic and neurological pathologies, who undergo rehabilitation at the FPG Hospitalization and Rehabilitation Services clinic.
Sampling Method: Probability Sample
Enrollment: 23 (Estimated)
Dates: Start 2022-02-17 (Actual); Primary Completion 2024-02-17 (Estimated); Study Completion 2024-02-17 (Estimated)

PRIMARY OUTCOMES:
Cobb angle | This is a baseline evaluation. The study does not include further evaluations. We aimed to perform a one-time comparison of the Cobb's angle measured through BHOHB SPINAL-METER versus standard spinal radiography
  radiographic angle measuring the degree of scoliosis in the frontal plane

SECONDARY OUTCOMES:
Berg Balance scale | This is a baseline evaluation. The study does not include further evaluations. The Berg balance scale score goes from 0 to 56 points. Higher scores indicate low/no balance deficit and low/no risk of falling.
  balance scale
Tinetti scale | This is a baseline evaluation. The study does not include further evaluations. The Tinetti scale score goes from 0 to 26. The higher scores indicate a lower risk of falls
  balance and deambulation scale
NRS numeric rating scale for pain | This is a baseline evaluation. The study does not include further evaluations. NRS score goes from 0 to 10. Higher scores correspond to worse pain perception.
  visual analogical scale for pain assessment
stabilometric test | This is a baseline evaluation. The study does not include further evaluations.
  assessment of static balance

CONTACTS AND LOCATIONS:
Overall Officials: gianpaolo ronconi, Principal Investigator — Catholic University of the Sacred Heart
Locations (1):
- Gianpaolo Ronconi, Roma, Italy

REFERENCES:
- [Background] Tinetti ME. Performance-oriented assessment of mobility problems in elderly patients. J Am Geriatr Soc. 1986 Feb;34(2):119-26. doi: 10.1111/j.1532-5415.1986.tb05480.x. No abstract available. PMID 3944402
- [Background] Berg KO, Wood-Dauphinee SL, Williams JI, Maki B. Measuring balance in the elderly: validation of an instrument. Can J Public Health. 1992 Jul-Aug;83 Suppl 2:S7-11. PMID 1468055
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Cohen L, Kobayashi S, Simic M, Dennis S, Refshauge K, Pappas E. Non-radiographic methods of measuring global sagittal balance: a systematic review. Scoliosis Spinal Disord. 2017 Oct 3;12:30. doi: 10.1186/s13013-017-0135-x. eCollection 2017. PMID 29026895